CLINICAL TRIAL: NCT01120314
Title: An Open-label Pharmacokinetic, Pharmacodynamic and Tolerability Study of Otamixaban Given as a Single 80 μg/kg Bolus Plus 100 µg/kg/h Continuous Infusion for 24 Hours in Subjects With Mild, Moderate and Severe Renal Impairment, and in Matched Subjects With Normal Renal Function
Brief Title: Pharmacokinetic, Pharmacodynamic and Tolerability Study of Otamixaban in Patients With Mild, Moderate and Severe Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: POP6537; U1111-1116-5821 (Other: UTN)
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Renal Impairment
MeSH Terms: conditions — Renal Insufficiency | interventions — otamixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Severe renal impairment population (Experimental)
  Interventions: Drug: OTAMIXABAN (XRP0673)
- Moderate renal impairment population (Experimental)
  Interventions: Drug: OTAMIXABAN (XRP0673)
- Mild renal impairment population (Experimental)
  Interventions: Drug: OTAMIXABAN (XRP0673)
- Healthy population (Experimental): Healthy matched subjects
  Interventions: Drug: OTAMIXABAN (XRP0673)

INTERVENTIONS:
Drug: OTAMIXABAN (XRP0673) — Form: solution for injection
  Route: intravenous

SUMMARY:
Primary Objective:

* To study effect of mild, moderate and severe renal impairment on the pharmacokinetics of Otamixaban.

Secondary Objective:

* To assess the pharmacodynamic effects of Otamixaban on subjects with mild, moderate and severe renal impairment and in matched subjects with normal renal function.

DETAILED DESCRIPTION:
The study period for one subject is broken down as follows:

* 2 to 28 days of screening,
* 1 day of treatment,
* 8 to 11 days of follow-up after start of infusion.

There are 5 days in the unit starting the day before the start of infusion.

ELIGIBILITY:
Inclusion criteria:

* Subject with renal impairment:

  * Mild, moderate or severe renal impairment defined as Creatinine Clearance (CrCl) from 50 to 80, 30 to 50 and < 30 mL/min respectively, based on the Cockcroft-Gault formula,
  * Body weight between 50.0 kg and 115.0 kg inclusive if male, between 40.0 kg and 95.0 kg inclusive if female, Body Mass Index between 18.0 and 34.9 kg/m2 inclusive.
  * Stable chronic renal impairment as defined by Cockcroft-Gault formula,
  * Vital signs, cardiac function and laboratory parameters within the acceptable range.
* Or matched subject (by age, gender and body weight) with normal renal function (defined as CrCl >80 mL/min) and certified as healthy by physical examination, medical history and laboratory findings.
* If female, subject must use a double contraception method, except if she is sterilized for more than 3 months or postmenopausal.

Exclusion criteria:

* Uncontrolled clinically relevant cardiovascular, pulmonary, gastro-intestinal, metabolic, hematological, neurological, psychiatric, systemic, ocular, gynecologic (if female) or infectious disease, or signs of acute illness.
* Active hepatitis, hepatic insufficiency.
* Acute renal failure, nephrotic syndrome.
* History of or current hematuria of urologic origin.
* Subject requiring dialysis during the study.
* History or presence of drug or alcohol abuse within two years before inclusion.
* Smoking more than 15 cigarettes or equivalent per day.
* Any significant change in chronic treatment medication within 14-days before inclusion.

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2010-04; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of Otamixaban (Observed concentration at the end of the infusion (Ceoi) and Areas Under the plasma concentration Curve(AUClast and AUC)) | 4 days

SECONDARY OUTCOMES:
Pharmacodynamic effect based on coagulation parameters (activated Partial Prothrombin Time (aPTT), Prothrombin Time (PT) and International Normalized Ratio (INR)) | 4 days

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (4):
- United States (4):
  - Investigational Site Number 840003, Miami Gardens, Florida
  - Investigational Site Number 840005, Orlando, Florida
  - Investigational Site Number 840004, Saint Paul, Minnesota
  - Investigational Site Number 840002, Knoxville, Tennessee